CLINICAL TRIAL: NCT06926153
Title: Evaluation of an Intervention to Reduce Smoking Among Mental Health Users Treated in Ambulatory Psychiatry
Brief Title: Interventional Study on Smoking Reduction in Psychiatry
Acronym: TABAPSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS-CCOMS (Other)
Collaborators: INSERM ECEVE 1123 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A01474-43; A19017HS (Other: Institute for Public Health Research (IRESP))
Record Dates: First submitted 2025-02-18; First posted 2025-04-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Addiction
Keywords: Smoking reduction; People with mental disorders; Psychiatry
MeSH Terms: conditions — Smoking Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Sectors randomized to the intervention group will implement the 'Tabapsy' intervention.
  Interventions: Other: TABAPSY
- Usual care (Other): Sectors randomized to the control group will continue implementing their usual smoking cessation promotion.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: TABAPSY — The Tabapsy intervention consists in a campaign to promote smoking cessation within the CMP, and an intervention to help people stop smoking which comprises of a) A general information meeting; b) An assessment workshop, to evaluate level of dependence using validated tests and establish a personalized cessation program based on the results obtained; c) Five thematic workshops to support cessation, covering 1/ nicotine replacement treatments, electronic cigarettes and other drug treatments available for smoking cessation, 2/ emotional management, 3/ weight gain, 4/ physical activities, and 5/ manual occupations; d) Peer support groups, based on the sharing of experiences, to encourage mutual aid and solidarity between people with mental disorders who are trying to quit smoking.
  The intervention relies on a facilitator specifically recruited to implement and run the intervention in the CMP. It is complemented by a website that will contain all the resources and information presented dur
  Arms: Intervention arm
Other: Usual Care — Usual care corresponds to usual practices regarding smoking cessation activities in participating sectors. Those practices may vary (enquiring whether a patient is a smoker or not, offering smoking cessation if they are or only if the patient asks, etc.)
  Arms: Usual care

SUMMARY:
The smoking rate among people with mental disorders is higher than in the general population. Greater exposure to the harmful effects of tobacco partly explains the major inequality in life expectancy observed among people with mental disorders who, depending on the disorder and the study, live 10 to 25 years less than the general population, a gap mainly due to the occurrence of cardiovascular and respiratory pathologies, notably bronchial cancers. However, tobacco reduction actions specifically targeting these people remain insufficiently developed, particularly in psychiatry where this addiction is often banalized and its treatment neglected.

The objective of this study is to evaluate an intervention ('Tabapsy') co-constructed with mental health services users, mental health professionals, and general practitioners and targeting adult patients followed in ambulatory psychiatry. The main objective is to evaluate the effectiveness of the intervention on short-term smoking cessation (cessation for at least 7 days) among regular smokers at 3 months. Secondary objectives include evaluation of its cost-effectiveness and implementation. To this end, a national cluster-randomized controlled study will be carried out, supplemented by qualitative interviews to study the implementation of the intervention.

DETAILED DESCRIPTION:
The smoking rate among people with mental disorders is higher than in the general population. Greater exposure to the harmful effects of tobacco partly explains the major inequality in life expectancy observed among people with mental disorders who, depending on the disorder and the study, live 10 to 20 years less than the general population, a gap mainly due to the occurrence of cardiovascular and respiratory pathologies, notably bronchial cancers.

While studies found that people under psychiatric care are as motivated as others to stop smoking, the literature also shows that psychiatric care systems tolerate, underestimate and even encourage smoking among users, despite the fact that psychiatric care, whether at hospital or in an ambulatory setting, is conducive to changes in smoking behaviour and to the implementation of a smoking cessation approach, notably because of anti-smoking regulations in hospitals. In addition, withdrawal symptoms is stronger in this population and smoking cessation would therefore need to be adapted.

Against this backdrop, a smoking cessation intervention ('Tabapsy') was co-constructed with the various stakeholders (users with mental disorders, mental health professionals and general practitioners). Its aim is to encourage and support smoking cessation among people with mental disorders followed in ambulatory psychiatry by medical psychological centers (CMP). It consists of two parts: a campaign to promote smoking cessation within the CMP, and the setting up of an intervention to help people stop smoking. The latter comprises of:

1. A general information meeting, to encourage motivation to start smoking cessation;
2. An assessment workshop, to evaluate level of dependence using validated tests and establish a personalized cessation program based on the results obtained;
3. Five thematic workshops to support cessation, covering 1/ nicotine replacement treatments, electronic cigarettes and other drug treatments available for smoking cessation, 2/ emotional management, 3/ weight gain, 4/ physical activities, and 5/ manual occupations;
4. Peer support groups, based on the sharing of experiences, to encourage mutual aid and solidarity between people with mental disorders who are trying to quit smoking.

The intervention also relies on a facilitator specifically recruited to set up the intervention and run the various workshops in the CMP. It is complemented by a website that will contain all the resources and information presented during the meetings/workshops.

The primary objective of the study is to evaluate the effectiveness of the "Tabapsy" intervention on short-term smoking cessation (cessation for at least 7 days) at 3 months among regular smokers followed by adult psychiatric CMPs. Secondary objectives include assessing its cost-effectiveness and implementation.

A cluster-randomized controlled trial will be carried out to evaluate the intervention. The cluster is the "psychiatric sector", i.e., the public care entity responsible for organizing the mental health care of a population within a pre-specified geographical area (including hospital and ambulatory care) in France. A psychiatric sector may include one or multiple CMPs depending on the size of the population it serves. Psychiatric sectors will be randomized into one of two groups (intervention or usual practice).

It will be supplemented by a qualitative study to study the implementation of the intervention.

All regular smokers (at least one cigarette a day) who agree to participate will be asked to complete questionnaires on a WebApp at inclusion, and again at 3 and 6 months. Additional questionnaires will be available in the intervention group. Questions will focus on user characteristics, tobacco consumption, level of nicotine dependence, motivation to quit, use of cessation aids, level of mental and physical well-being, smoking-related knowledge and representations, and in the intervention group, participation in the intervention and satisfaction.

6,250 participants will be included over 12 months, in 22 participating sectors.

ELIGIBILITY:
Inclusion Criteria:

* Regular smokers (at least one cigarette per day)
* Followed in psychiatric ambulatory care at one of the participating sectors' CMPs
* Adults (18 years or older)
* Covered by the statuary health insurance
* Who gave their informed consent to participate to the study

Exclusion Criteria:

* Users under guardianship or legal protection,
* Psychological state incompatible with completing the questionnaire,
* Persons with no command or understanding of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6500 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Short-term smoking cessation | 3 months
  Short-term smoking cessation corresponds to a smoking cessation of at least 7 days, assessed among regular smoker (at least one cigarette a day) included in the study.

SECONDARY OUTCOMES:
Motivation to stop smoking | 3 and 6 months
  The motivation to stop smoking will be assessed using the Q-Mat ("Questionnaire de motivation à l'arrêt du tabac") scale. The computed score ranges from 0 to 20, 20 representing the highest motivation.
Voluntary quit attempts lasting at least 24 hours in the last 3 months | 3 and 6 months
  Number of voluntary quit attempts assessed both as percentage of users reporting at least one quit attempt and mean number of quit attempts per use
Voluntary quit attempts lasting at least 7 days in the last 3 months | 3 and 6 months
  Number of voluntary quit attempts assessed both as percentage of users reporting at least one quit attempt and mean number of quit attempts per user.
Tobacco consumption | 3 and 6 months
  Number of cigarettes smoked per day
Nicotine dependence | 3 and 6 months
  Nicotine dependence will be measured by the 6-question Fagerström test.
Short-term smoking cessation | 6 months
  Short-term smoking cessation corresponds to a smoking cessation of at least 7 days, assessed among regular smoker (at least one cigarette a day) included in the study.
Medium-term smoking cessation | At 3 and 6 months
  Medium-term smoking cessation corresponds to a smoking cessation of at least 30 days, assessed among regular smoker (at least one cigarette a day) included in the study.
Use of smoking cessation aids | 3 and 6 months
  Number of participants using smoking cessation aids (nicotine replacement therapy and other smoking cessation medications (varenicline or bupropion), electronic cigarettes, and health professionals, assessed together and separately
Level of mental well-being | 3 and 6 months
  Level of mental well-being assessed with a visual analog scale ranging from 1 to 10, 10 representing the highest level of mental well-being
Level of physical well-being | 3 and 6 months
  Level of physical well-being assessed with a visual analog scale ranging from 1 to 10, 10 representing the highest level of physical well-being
Knowledge and representations surrounding tobacco use | 3 and 6 months
  Knowledge and representations surrounding tobacco use will be assessed using a dedicated questionnaire addressed to all the included population as well as to patients who participated to a given workshop
Cost-effectiveness (short-term) | A 6 months
  Incremental cost-effectiveness ratio in cost per additional weaning of at least 7 days.
Cost-effectiveness (long-term) | 6 months
  Incremental cost-effectiveness ratio in cost per life-year gained over the entire life of users, using extrapolated data and economic modeling (Markov model) to assess lifetime costs and effectiveness 'till all patients in the model are deceased.
Budgetary impact (costs) | 5 years after hypothetical generalization
  Direct costs will be calculated with and without the Tabapsy intervention to assess the budgetary impact of its generalization.
Budgetary impact (health benefits) | 5 years after hypothetical generalization
  The number of users who have stopped smoking for at least 7 days will be calculated with and without the Tabapsy intervention to assess the health gains associated with its generalization.
Implementation | 6 months
  The implementation of the intervention and its components will be assessed using qualitative methods through semi-structured interviews conducted with 25 mental health users et 25 mental health professionnals of the intervention group).
Satisfaction level | 3 and 6 months
  Users who participated in one of the components of the intervention will be asked to rate their satisfaction using a visual analog scale ranging from 0 to 10, with 10 corresponding to the highest satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc ROELANDT, MD, Principal Investigator — GCS-CCOMS & INSERM ECEVE 1123; Karine CHEVREUL, MD and Pr of public health, Study Director — Evaluation and research in health services and policies for vulnerable populations, French National Institute for Health and Medical Research (INSERM ECEVE 11 23)
Locations (22):
- France (19):
  - Public mental health establishment of Lille Metropole (59G16-G17), Armentières
  - Public mental health establishment of Lille Metropole (59G21), Armentières
  - Flanders public mental health establishment (59G05/06), Bailleul
  - Barthelemy Durand public health establishment (91G05), Étampes
  - Psychotherapeutic center of Nancy (54G02-06), Laxou
  - University Hospital Center of Lille (59G08), Lille
  - Hospital Care Center of Nanterre (92G10), Nanterre
  - University Hospital Group Paris Neurosciences & Psychiatry (75G04), Paris
  - Hospital Center of Rouffach (68G02/03), Rouffach
  - Hospital Center of Rouffach (68G08/09), Rouffach
  - Hospital Center of Rouffach (Pôle LTD - 68G04/05), Rouffach
  - Hospitals of Paris Est Val de Marne (94G01), Saint-Maurice
  - Hospitals of Paris Est Val de Marne (94G16), Saint-Maurice
  - Hospitals of Paris Est Val de Marne (Paris 11), Saint-Maurice
  - Hospitals of Paris Est Val de Marne (Paris 12), Saint-Maurice
  - Hospitals of Paris Est Val de Marne (Paris Centre), Saint-Maurice
  - Public mental health establishment of Val de Lys Artois (62G09), Saint-Venant
  - Public mental health establishment of Val de Lys Artois (62G12), Saint-Venant
  - Public mental health establishment of Val de Lys Artois (Pôle du Ternois), Saint-Venant
- Guadeloupe (2):
  - Public mental health establishment of Guadeloupe (96G01), Saint-Claude
  - Public mental health establishment of Guadeloupe (96G06), Saint-Claude
- Public mental health establishment of Reunion Island (Pôle Nord), Saint-Paul, Reunion

IPD SHARING:
Plan to Share IPD: No